CLINICAL TRIAL: NCT03090217
Title: Pelvic Physiotherapy in the Prevention of Vaginal Stenosis Secondary to Radiotherapy of Gynecological Cancer: a Randomized Controlled Trial
Brief Title: Pelvic Physiotherapy in the Prevention of Vaginal Stenosis Secondary to the Radiotherapy
Acronym: PPPVSSR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PP-radiotherapy 2017
Record Dates: First submitted 2017-01-12; First posted 2017-03-24 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Gynecologic Cancer; Pathological Constriction
Keywords: Radiotherapy; Brachytherapy; Physiotherapy; Vaginal dilators; Pelvic floor exercises; Vaginal Stenosis
MeSH Terms: conditions — Constriction, Pathologic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic physiotherapy (PP) (Experimental): Pelvic Physiotherapy include daily pelvic floor muscle training (PFMT). PFMT starts at first session of the brachytherapy and will be conduced during the twelve weeks treatment.
  Interventions: Behavioral: Pelvic Physiotherapy; Behavioral: Standard care (SC)
- Stander Care (SC) (Active Comparator): The stander care (SC) includes a guideline for gynecological cancer patients under radiotherapy/brachytherapy: 1) daily vaginal dilator therapy (10 to 15 minutes); and 2) usual care management. This SC starts at first session of the brachytherapy and will be conduced during the twelve weeks treatment.
  Interventions: Behavioral: Standard care (SC)

INTERVENTIONS:
Behavioral: Pelvic Physiotherapy — 1) daily pelvic floor muscle training (PFMT).
  Other Names: PFMT
  Arms: Pelvic physiotherapy (PP)
Behavioral: Standard care (SC) — 1) daily vaginal dilator therapy (10 to 15 minutes) and 2) usual care management.
  Other Names: SC

SUMMARY:
Vaginal stenosis is one of the most prevalent side effects of pelvic radiation, affecting about one third of women. In this randomized controlled trial, the effect of a pelvic physiotherapy protocol on an incidence rate of vaginal stenosis in women with gynecological cancer undergoing gynecological brachytherapy. In addition, the investigators will explore an improvement in quality of life, sexuality, and contractile function of the pelvic floor muscles.

DETAILED DESCRIPTION:
Tis study will be conducing in a reference hospital to oncology treatment were mane patients with gynecologic cancer are management on radiotherapy services. The aim of this work is evaluated the effects of the pelvic physiotherapy (PP) on the more prevalent constriction pathology (vaginal stenosis) secondary to the brachytherapy. The PP will be conduced by three months after the radiotherapy starts and the incidence of the vaginal stenosis will be compared with a control group throughout six months of fallow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old;
* No vaginal stenosis at first evaluation;
* Women free of previous intracavitary radiation;
* Women diagnosed with gynecological cancer who are undergoing brachytherapy treatment during the period of research at the Santa Rita Hospital of the Santa Casa de Misericórdia in Porto Alegre;
* Women who agree to participate in the research through the Informed Consent Form (TCLE).

Exclusion Criteria:

* Women who do not sign the ICF;
* Women not being treated for gynecological cancer;
* Women who have a 30% lack of physical therapy sessions (4 sessions);
* Women who present complications that prevent the accomplishment of the protocol of pelvic physiotherapy or that do not perform all the treatment with brachytherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-08-21 (Estimated); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal Stenosis | With completion of the study, predicted 15 months after the start of the study.
  Vaginal stenosis will be evaluated before the first brachytherapy and twelve months after. Considered according to the study of Kirchheiner et al., (2016) that used the Common Terminology Criteria for Adverse Events (CTCAE v3.0). Vaginal stenosis will also be considered as the narrowing of the vaginal canal that makes it impossible to introduce the number 1 acrylic gynecological speculum through the vaginal introitus.

SECONDARY OUTCOMES:
Quality of life | With completion of the study, predicted 15 months after the start of the study.
  The quality of live will be evaluated before the first brachytherapy and twelve months after through the application of the Quality of Life questionnaire European Organization for Research and Treatment of Cancer - EORTC QLQ-C30.
Sexuality | With completion of the study, predicted 15 months after the start of the study.
  The sexuality will be evaluated before the first brachytherapy and twelve months after through the application of the questionnaire The Female Sexual Function Index (FSFI).
Muscle activity and contractile function of the pelvic floor | With completion of the study, predicted 15 months after the start of the study.
  Measurement of pelvic floor activity will be evaluated before the first brachytherapy and twelve months after through surface electromyography (EMG), which is able to record the extracellular bioelectric activity generated by muscle fibers, through the electromyographic biofeedback Miotool 400 from Miotec.

OTHER OUTCOMES:
The vaginal area | With completion of the study, predicted 15 months after the start of the study.
  The vaginal area will be evaluated before the first brachytherapy and twelve months after through A-SÒS-labeled vaginal dilators in eight different sizes in square centimeters and the vaginal length will be measured with a hysterometer, introduced into the vaginal canal until it reaches the cervix (from the himenal ring to the Posterior fornice), the measurement will be in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Taís M Cerentini, Bela., Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Comitê de Ética em Pesquisa - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
If shared, available after the end of the study through email taismcerentini@gmail.com

REFERENCES:
- [Background] ABHINAV, KR et al. Analysis of Late Radiation Proctitis Among Patients Treated for Cervical Cancer: A Comparative Study Between Linear Accelerator and Cobalt Teletherapy. Clinical Ovarian and Other Gynecologic Cancer, 6(1): 46-49, 2013.
- [Background] Auchincloss CC, McLean L. The reliability of surface EMG recorded from the pelvic floor muscles. J Neurosci Methods. 2009 Aug 30;182(1):85-96. doi: 10.1016/j.jneumeth.2009.05.027. Epub 2009 Jun 17. PMID 19539646
- [Background] Bahng AY, Dagan A, Bruner DW, Lin LL. Determination of prognostic factors for vaginal mucosal toxicity associated with intravaginal high-dose rate brachytherapy in patients with endometrial cancer. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):667-73. doi: 10.1016/j.ijrobp.2010.10.071. Epub 2011 Feb 6. PMID 21300451
- [Background] Bakker RM, Vermeer WM, Creutzberg CL, Mens JW, Nout RA, Ter Kuile MM. Qualitative accounts of patients' determinants of vaginal dilator use after pelvic radiotherapy. J Sex Med. 2015 Mar;12(3):764-73. doi: 10.1111/jsm.12776. Epub 2014 Nov 25. PMID 25424559
- [Background] Bernards AT, Berghmans BC, Slieker-Ten Hove MC, Staal JB, de Bie RA, Hendriks EJ. Dutch guidelines for physiotherapy in patients with stress urinary incontinence: an update. Int Urogynecol J. 2014 Feb;25(2):171-9. doi: 10.1007/s00192-013-2219-3. Epub 2013 Oct 1. PMID 24081496
- [Background] BERNARDO, BC et al. Disfunção sexual em pacientes com câncer do colo uterino avançado submetidas à radioterapia exclusiva. Revista Brasileira de Ginecologia e Obstetrícia, 29(2): 85-90, 2007.
- [Background] Bi X, Zhao J, Zhao L, Liu Z, Zhang J, Sun D, Song L, Xia Y. Pelvic floor muscle exercise for chronic low back pain. J Int Med Res. 2013 Feb;41(1):146-52. doi: 10.1177/0300060513475383. Epub 2013 Jan 23. PMID 23569140
- [Background] Brand AH, Bull CA, Cakir B. Vaginal stenosis in patients treated with radiotherapy for carcinoma of the cervix. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):288-93. doi: 10.1111/j.1525-1438.2006.00348.x. PMID 16445647
- [Background] Brand AH, Do V, Stenlake A. Can an educational intervention improve compliance with vaginal dilator use in patients treated with radiation for a gynecological malignancy? Int J Gynecol Cancer. 2012 Jun;22(5):897-904. doi: 10.1097/IGC.0b013e31824d7243. PMID 22552831
- [Background] BO, K et al. Pelvic floor muscle exercise for the treatment of female stress urinary incontinence: II. Validity of vaginal pressure measurements of pelvic floor muscle strength and the necessity of supplementary methods for control of correct contraction. Neurourology and Urodynamics, 9(5): 479-487, 1990.
- [Background] Bruner DW, Lanciano R, Keegan M, Corn B, Martin E, Hanks GE. Vaginal stenosis and sexual function following intracavitary radiation for the treatment of cervical and endometrial carcinoma. Int J Radiat Oncol Biol Phys. 1993 Nov 15;27(4):825-30. doi: 10.1016/0360-3016(93)90455-5. PMID 8244811
- [Background] Bruner DW, Nolte SA, Shahin MS, Huang HQ, Sobel E, Gallup D, Cella D; Gynecologic Oncology Group. Measurement of vaginal length: Reliability of the vaginal sound--a Gynecologic Oncology Group study. Int J Gynecol Cancer. 2006 Sep-Oct;16(5):1749-55. doi: 10.1111/j.1525-1438.2006.00711.x. PMID 17009966
- [Background] CANTEIRO, R. Avaliação do comprimento da cavidade uterina por meio da histerometria e ultrassom em mulheres nuligestas e com gestação prévia. 2009. 56 p. Dissertação de Mestrado para obtenção do grau Mestre em Tocoginecologia, área de Ciências Biomédicas.Campinas, SP. 2009.
- [Background] Carpenter JS, Reed SD, Guthrie KA, Larson JC, Newton KM, Lau RJ, Learman LA, Shifren JL. Using an FSDS-R Item to Screen for Sexually Related Distress: A MsFLASH Analysis. Sex Med. 2015 Mar;3(1):7-13. doi: 10.1002/sm2.53. PMID 25844170
- [Background] Carter J, Goldfrank D, Schover LR. Simple strategies for vaginal health promotion in cancer survivors. J Sex Med. 2011 Feb;8(2):549-59. doi: 10.1111/j.1743-6109.2010.01988.x. Epub 2010 Aug 16. PMID 20722792
- [Background] CICONELLI, RM. Tradução para o português e validação do questionário genérico de avaliação de qualidade de vida Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). Revista Brasileira de Reumatologia. 39(3), 1999.
- [Background] Nascimento-Correia G, Santos-Pereira V, Tahara N, Driusso P. [Effects of pelvic floor muscle training on quality of life of a group of women with urinary incontinence: randomized controlled trial]. Actas Urol Esp. 2012 Apr;36(4):216-21. doi: 10.1016/j.acuro.2011.07.007. Epub 2011 Sep 28. Spanish. PMID 21959066
- [Background] Cullen K, Fergus K, Dasgupta T, Fitch M, Doyle C, Adams L. From "sex toy" to intrusive imposition: a qualitative examination of women's experiences with vaginal dilator use following treatment for gynecological cancer. J Sex Med. 2012 Apr;9(4):1162-73. doi: 10.1111/j.1743-6109.2011.02639.x. Epub 2012 Feb 3. PMID 22304701
- [Background] Cullen K, Fergus K, DasGupta T, Kong I, Fitch M, Doyle C, Adams L. Toward clinical care guidelines for supporting rehabilitative vaginal dilator use with women recovering from cervical cancer. Support Care Cancer. 2013 Jul;21(7):1911-7. doi: 10.1007/s00520-013-1726-6. Epub 2013 Feb 17. PMID 23417563
- [Background] Decruze SB, Guthrie D, Magnani R. Prevention of vaginal stenosis in patients following vaginal brachytherapy. Clin Oncol (R Coll Radiol). 1999;11(1):46-8. doi: 10.1053/clon.1999.9008. PMID 10194586
- [Background] Denton AS, Maher EJ. Interventions for the physical aspects of sexual dysfunction in women following pelvic radiotherapy. Cochrane Database Syst Rev. 2003;2003(1):CD003750. doi: 10.1002/14651858.CD003750. PMID 12535485
- [Background] Faubion SS, MacLaughlin KL, Long ME, Pruthi S, Casey PM. Surveillance and Care of the Gynecologic Cancer Survivor. J Womens Health (Larchmt). 2015 Nov;24(11):899-906. doi: 10.1089/jwh.2014.5127. Epub 2015 Jul 24. PMID 26208166
- [Background] Flay LD, Matthews JH. The effects of radiotherapy and surgery on the sexual function of women treated for cervical cancer. Int J Radiat Oncol Biol Phys. 1995 Jan 15;31(2):399-404. doi: 10.1016/0360-3016(94)E0139-B. PMID 7836095
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Franceschini J, Jardim JR, Fernandes AL, Jamnik S, Santoro IL. Reproducibility of the Brazilian Portuguese version of the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire used in conjunction with its lung cancer-specific module. J Bras Pneumol. 2010 Sep-Oct;36(5):595-602. doi: 10.1590/s1806-37132010000500011. English, Portuguese. PMID 21085825
- [Background] FRIGATO, S; HOGA, LAK. Assistência à mulher com câncer de colo uterino: o papel da enfermagem. Rev Bras Cancerol, 49(4): 209-14, 2003.
- [Background] Grape HH, Dedering A, Jonasson AF. Retest reliability of surface electromyography on the pelvic floor muscles. Neurourol Urodyn. 2009;28(5):395-9. doi: 10.1002/nau.20648. PMID 19214991
- [Background] Grion RC, Baccaro LF, Vaz AF, Costa-Paiva L, Conde DM, Pinto-Neto AM. Sexual function and quality of life in women with cervical cancer before radiotherapy: a pilot study. Arch Gynecol Obstet. 2016 Apr;293(4):879-86. doi: 10.1007/s00404-015-3874-z. Epub 2015 Aug 29. PMID 26319157
- [Background] Hata M, Koike I, Miyagi E, Numazaki R, Asai-Sato M, Kasuya T, Kaizu H, Matsui T, Hirahara F, Inoue T. Radiation therapy for pelvic lymph node metastasis from uterine cervical cancer. Gynecol Oncol. 2013 Oct;131(1):99-102. doi: 10.1016/j.ygyno.2013.07.085. Epub 2013 Jul 19. PMID 23877014
- [Background] HENTSCHEL, H et al. Validação do Female Sexual Function Index (FSFI) para uso em língua portuguesa. Rev HCPA, 27(1): 10-4, 2007.
- [Background] Huang Z, Zheng Y, Wen W, Wu C, Bao P, Wang C, Zhong W, Gao YT, Jin F, Xiang YB, Shu XO, Beeghly-Fadiel A. Incidence and mortality of gynaecological cancers: Secular trends in urban Shanghai, China over 40 years. Eur J Cancer. 2016 Aug;63:1-10. doi: 10.1016/j.ejca.2016.04.016. Epub 2016 May 26. PMID 27254837
- [Background] Instituto Nacional de Câncer. Tipos de câncer. Disponível em: <http://www2.inca.gov.br/wps/wcm/connect/tiposdecancer/site/home/colo_utero/definicao>. Acesso em: 30.ago.2016.
- [Background] Instituto Nacional de Câncer. Câncer do colo do útero. Disponível em: http://www.inca.gov.br/estimativa/2016/sintese-de-resultados-comentarios.asp. Acesso em 19.set.2016.
- [Background] KEGEL AH. Progressive resistance exercise in the functional restoration of the perineal muscles. Am J Obstet Gynecol. 1948 Aug;56(2):238-48. doi: 10.1016/0002-9378(48)90266-x. No abstract available. PMID 18877152
- [Background] Kirchheiner K, Nout RA, Lindegaard JC, Haie-Meder C, Mahantshetty U, Segedin B, Jurgenliemk-Schulz IM, Hoskin PJ, Rai B, Dorr W, Kirisits C, Bentzen SM, Potter R, Tanderup K; EMBRACE Collaborative Group. Dose-effect relationship and risk factors for vaginal stenosis after definitive radio(chemo)therapy with image-guided brachytherapy for locally advanced cervical cancer in the EMBRACE study. Radiother Oncol. 2016 Jan;118(1):160-6. doi: 10.1016/j.radonc.2015.12.025. Epub 2016 Jan 9. PMID 26780997
- [Background] Knorst MR, Resende TL, Santos TG, Goldim JR. The effect of outpatient physical therapy intervention on pelvic floor muscles in women with urinary incontinence. Braz J Phys Ther. 2013 Sep-Oct;17(5):442-9. doi: 10.1590/S1413-35552012005000117. Epub 2013 Oct 21. English, Portuguese. PMID 24173346
- [Background] Lancaster L. Preventing vaginal stenosis after brachytherapy for gynaecological cancer: an overview of Australian practices. Eur J Oncol Nurs. 2004 Mar;8(1):30-9. doi: 10.1016/S1462-3889(03)00059-0. PMID 15003742
- [Background] LATORRE, GFS et al. Escores de corte para o FSFI. Revista Inspirar Movimento & Saude, 7(1), 2015.
- [Background] Law E, Kelvin JF, Thom B, Riedel E, Tom A, Carter J, Alektiar KM, Goodman KA. Prospective study of vaginal dilator use adherence and efficacy following radiotherapy. Radiother Oncol. 2015 Jul;116(1):149-55. doi: 10.1016/j.radonc.2015.06.018. Epub 2015 Jul 8. PMID 26164775
- [Background] Mahmud A, Brydon B, Tonita J, Hanna TP, Schmidt M, Tai P. A population-based study of cervix cancer: incidence, management and outcome in the Canadian province of Saskatchewan. Clin Oncol (R Coll Radiol). 2011 Dec;23(10):691-5. doi: 10.1016/j.clon.2011.05.002. Epub 2011 Jun 8. PMID 21646003
- [Background] MENEZES, AMB; SANTOS, IS. Curso de epidemiologia básica para pneumologistas. Jornal Brasileiro de Pneumologia, 25(3): 163-166, 1999.
- [Background] Miles T, Johnson N. Vaginal dilator therapy for women receiving pelvic radiotherapy. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007291. doi: 10.1002/14651858.CD007291.pub2. PMID 20824858
- [Background] Mohamed S, Lindegaard JC, de Leeuw AA, Jurgenliemk-Schulz I, Kirchheiner K, Kirisits C, Potter R, Tanderup K. Vaginal dose de-escalation in image guided adaptive brachytherapy for locally advanced cervical cancer. Radiother Oncol. 2016 Sep;120(3):480-485. doi: 10.1016/j.radonc.2016.05.020. Epub 2016 Jun 3. PMID 27267048
- [Background] MORENO, A. Fisioterapia em Uroginecologia, Avaliação Fisioterapêutica, 1:101-112, 2004.
- [Background] Nunns D, Williamson K, Swaney L, Davy M. The morbidity of surgery and adjuvant radiotherapy in the management of endometrial carcinoma. Int J Gynecol Cancer. 2000 May;10(3):233-238. doi: 10.1046/j.1525-1438.2000.010003233.x. PMID 11240680
- [Background] Occhino JA, Trabuco EC, Heisler CA, Klingele CJ, Gebhart JB. Changes in vaginal anatomy and sexual function after vaginal surgery. Int Urogynecol J. 2011 Jul;22(7):799-804. doi: 10.1007/s00192-011-1386-3. Epub 2011 Mar 17. PMID 21416284
- [Background] Olson B, Gribble B, Dias J, Curryer C, Vo K, Kowal P, Byles J. Cervical cancer screening programs and guidelines in low- and middle-income countries. Int J Gynaecol Obstet. 2016 Sep;134(3):239-46. doi: 10.1016/j.ijgo.2016.03.011. Epub 2016 May 26. PMID 27350227
- [Background] Organização Mundial de Saúde. Cadernos de atenção básica: controle dos cânceres do colo do útero e da mama. Brasilia: OMS, 2013. Ortiz OC, Coya NF, Ibanez G. Evaluación funcional del piso pelviano femenino (clasificación funcional). Soc Latinoam Uroginecol Cir Vaginal. 1996
- [Background] Park HS, Ratner ES, Lucarelli L, Polizzi S, Higgins SA, Damast S. Predictors of vaginal stenosis after intravaginal high-dose-rate brachytherapy for endometrial carcinoma. Brachytherapy. 2015 Jul-Aug;14(4):464-70. doi: 10.1016/j.brachy.2015.03.001. Epub 2015 Apr 14. PMID 25887343
- [Background] Phillips K, Hersch J, Turner R, Jansen J, McCaffery K. The influence of the 'cancer effect' on young women's responses to overdiagnosis in cervical screening. Patient Educ Couns. 2016 Oct;99(10):1568-75. doi: 10.1016/j.pec.2016.04.002. Epub 2016 Apr 16. PMID 27133918
- [Background] Polat M, Kahramanoglu I, Senol T, Senturk B, Ozkaya E, Karateke A. Comparison of the Effect of Laparoscopic and Abdominal Hysterectomy on Lower Urinary Tract Function, Vaginal Length, and Dyspareunia: A Randomized Clinical Trial. J Laparoendosc Adv Surg Tech A. 2016 Feb;26(2):116-21. doi: 10.1089/lap.2015.0437. Epub 2015 Dec 15. PMID 26671303
- [Background] Rakhra SS, Weaver C, Donnelly ED, Helenowski I, Prescott AE, Strauss JB. The effect of pelvic radiotherapy on vaginal brachytherapy cylinder diameter: Implications for optimal treatment order. Brachytherapy. 2016 Sep-Oct;15(5):549-53. doi: 10.1016/j.brachy.2016.04.391. Epub 2016 Jun 14. PMID 27317190
- [Background] ROSA, LM et al. Evaluation and classification of vaginal stenosis after brachytherapy. Texto & Contexto-Enfermagem, 25(2), 2016.
- [Background] Rosenbaum TY. Pelvic floor involvement in male and female sexual dysfunction and the role of pelvic floor rehabilitation in treatment: a literature review. J Sex Med. 2007 Jan;4(1):4-13. doi: 10.1111/j.1743-6109.2006.00393.x. PMID 17233772
- [Background] RESENDE, APM et al. Eletromiografia de superfície para avaliação dos músculos do assoalho pélvico feminino: revisão de literatura. Fisioterapia e Pesquisa, 2011
- [Background] Santa Mina D, Au D, Alibhai SM, Jamnicky L, Faghani N, Hilton WJ, Stefanyk LE, Ritvo P, Jones J, Elterman D, Fleshner NE, Finelli A, Singal RK, Trachtenberg J, Matthew AG. A pilot randomized trial of conventional versus advanced pelvic floor exercises to treat urinary incontinence after radical prostatectomy: a study protocol. BMC Urol. 2015 Sep 16;15:94. doi: 10.1186/s12894-015-0088-4. PMID 26377550
- [Background] Soares EM, Riul da Silva S. [Profile of patients with gynecological cancer under chemotherapy]. Rev Bras Enferm. 2010 Jul-Aug;63(4):517-22. doi: 10.1590/s0034-71672010000400003. Portuguese. PMID 20835653
- [Background] TAVARES, CMA; PRADO, ML. Pesquisando a prevenção do câncer ginecológico em Santa Catarina. Texto & contexto enferm, 15(4): 578-86, 2006.
- [Background] Thomas GM. Improved treatment for cervical cancer--concurrent chemotherapy and radiotherapy. N Engl J Med. 1999 Apr 15;340(15):1198-200. doi: 10.1056/NEJM199904153401509. No abstract available. PMID 10202172
- [Background] WOLF, JK. Prevention and treatment of vaginal stenosis resulting from pelvic radiation therapy. Community oncology, 3(10): 665-671, 2006
- [Background] Wright JJ, O'Connor KM. Female sexual dysfunction. Med Clin North Am. 2015 May;99(3):607-28. doi: 10.1016/j.mcna.2015.01.011. Epub 2015 Mar 6. PMID 25841603
- [Background] Yoshida K, Yamazaki H, Nakamura S, Masui K, Kotsuma T, Akiyama H, Tanaka E, Yoshikawa N, Uesugi Y, Shimbo T, Narumi Y, Yoshioka Y. Role of vaginal pallor reaction in predicting late vaginal stenosis after high-dose-rate brachytherapy in treatment-naive patients with cervical cancer. J Gynecol Oncol. 2015 Jul;26(3):179-84. doi: 10.3802/jgo.2015.26.3.179. Epub 2015 Apr 29. PMID 25925294
- [Background] Schover LR, Fife M, Gershenson DM. Sexual dysfunction and treatment for early stage cervical cancer. Cancer. 1989 Jan 1;63(1):204-12. doi: 10.1002/1097-0142(19890101)63:13.0.co;2-u. PMID 2910419
- [Background] Schvartzman R, Bertotto A, Schvartzman L, Wender MC. Pelvic floor muscle activity, quality of life, and sexual function in peri- and recently postmenopausal women with and without dyspareunia: a cross-sectional study. J Sex Marital Ther. 2014;40(5):367-78. doi: 10.1080/0092623X.2013.864363. Epub 2014 Jan 9. PMID 24279742
- [Background] VARTANIAN, JG et al. Questionários para a avaliação de qualidade de vida em pacientes com câncer de cabeça e pescoço validados no Brasil. Rev Bras Cir Cabeça Pescoço, 36(2): 108-15, 2007.
- [Background] Zomkowski K, Toryi AM, Sacomori C, Dias M, Sperandio FF. Sexual function and quality of life in gynecological cancer pre- and post-short-term brachytherapy: a prospective study. Arch Gynecol Obstet. 2016 Oct;294(4):833-40. doi: 10.1007/s00404-016-4099-5. Epub 2016 Apr 27. PMID 27117556
- [Derived] Cerentini TM, Schlottgen J, Viana da Rosa P, La Rosa VL, Vitale SG, Giampaolino P, Valenti G, Cianci S, Macagnan FE. Clinical and Psychological Outcomes of the Use of Vaginal Dilators After Gynaecological Brachytherapy: a Randomized Clinical Trial. Adv Ther. 2019 Aug;36(8):1936-1949. doi: 10.1007/s12325-019-01006-4. Epub 2019 Jun 17. PMID 31209699